CLINICAL TRIAL: NCT05186909
Title: A Randomized, Double-Blind, Placebo-Controlled Phase II Clinical Study to Evaluate the Efficacy and Safety of CM310 Recombinant Humanized Monoclonal Antibody Injection in Subjects With Moderate to Severe Asthma
Brief Title: A Study of CM310 in Subjects With Moderate to Severe Asthma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CM310-CSP-001
Record Dates: First submitted 2021-12-09; First posted 2022-01-11 (Actual); Last update posted 2024-02-28 (Actual); Status verified 2021-12

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- CM310 300mg Q2W (Experimental): CM310 is injected subcutaneously (SC) with a loading dose of 600 mg at the first dose, and then 300 mg each time, once every 2 weeks (Q2W) for a total of 12 doses.
  Interventions: Drug: CM310
- CM310 150mg Q2W (Experimental): CM310 is injected subcutaneously (SC) with a loading dose of 300 mg at the first dose, and then 150 mg each time, once every 2 weeks (Q2W) for a total of 12 doses.
  Interventions: Drug: CM310
- Placebo (Placebo Comparator): Subcutaneous injection (SC), once every 2 weeks (Q2W) for a total of 12 doses.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CM310 — CM310 Recombinant Humanized Monoclonal Antibody Injection
  Arms: CM310 150mg Q2W; CM310 300mg Q2W
Other: Placebo — Placebo
  Arms: Placebo

SUMMARY:
This study is a multi-center, randomized, double-blind, placebo-controlled Phase II clinical study to evaluate the efficacy, safety, PK characteristics, PD effects and immunogenicity of CM310 in subjects with moderate to severe asthma.

The study consists of three periods, including an up to 4-week screening period, a 24-week randomized treatment period, and a 8-week safety follow-up period.

ELIGIBILITY:
Inclusion Criteria:

* Subjects are able to understand the nature of the study and voluntarily sign the ICF.
* Diagnosed with asthma according to the 2021 version of the GINA guidelines for at least 1 year.
* Pre-bronchodilator FEV1 measurement ≤ 80% of predicted normal value.
* Subjects must have experienced a severe asthma exacerbation within 12 months prior to screening, and have not experienced a severe asthma exacerbation within 1 month prior to screening.

Exclusion Criteria:

* Women of childbearing potential have a positive pregnancy test result during the screening period; women who are pregnant or lactating.
* Received biologics with the same therapeutic purpose within 6 months prior to screening, such as similar IL-4Rα antagonist, IL-5/5R, anti-IgE monoclonal antibody (mAb).
* Diagnosed with chronic obstructive pulmonary disease (COPD) or other lung disorders that may compromise lung function (including but not limited to idiopathic pulmonary fibrosis, allergic granulomatous angiitis, bronchopulmonary aspergillosis allergic, pulmonary tuberculosis, etc.).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 52 (Actual)
Dates: Start 2022-01-12 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Change from baseline in pre-bronchodilator FEV1 (forced expiratory volume in 1 second) at 12 weeks. | 12 weeks
  Absolute change from baseline in pre-bronchodilator FEV1 in each dose group at 12 weeks of CM310 treatment compared with placebo.

SECONDARY OUTCOMES:
Change from baseline in pre-bronchodilator FEV1 at each evaluation time point. | 24 weeks
  Absolute change from baseline in pre-bronchodilator FEV1 at each evaluation time point.
Percent change from baseline in pre-bronchodilator FEV1 at each evaluation time point. | 24 weeks
  Percent change from baseline in pre-bronchodilator FEV1 at each evaluation time point.
Annualized rate of subjects experiencing severe asthma exacerbations. | 24 weeks
  Annualized rate of subjects experiencing severe asthma exacerbations during the 24-week randomized treatment period.
Time to the first onset of the severe asthma exacerbation event. | 24 weeks
  Time from baseline to the first onset of the severe asthma exacerbation event.
Annualized rate of subjects experiencing the event of loss of asthma control (LOAC). | 24 weeks
  Annualized rate of subjects experiencing the event of loss of asthma control (LOAC) during the 24-week randomized treatment period.
Time to the onset of the first event of LOAC. | 24 weeks
  Time from baseline to the onset of the first event of LOAC.
FEV1 percentage of predicted value (FEV1% Pred) | 32 weeks
  FEV1 percentage of predicted value (FEV1% Pred)
Peak diurnal and nocturnal expiratory flow (PEF) | 32 weeks
  Peak diurnal and nocturnal expiratory flow (PEF)
Forced vital capacity (FVC) | 32 weeks
  Forced vital capacity (FVC)
Maximal mid-expiratory flow (MMEF) | 32 weeks
  Maximal mid-expiratory flow (MMEF)
Change from baseline of FEV1 after the use of bronchodilator. | 32 weeks
  Change from baseline of FEV1 after the use of bronchodilator.
Change from baseline in the Asthma Control Questionnaire-5 (ACQ-5) score at each evaluation time point. | 32 weeks
  The ACQ-5 is a questionnaire used to evaluate the degree of asthma control. Each question is scored from 0 to 6 (on a 7-point scale) according to its severity. The higher the score, the less satisfactory symptom control is.
Change from baseline in asthma symptom score at each evaluation time point. | 32 weeks
  Patients will record total symptom scores in morning（a 0-4 scale, with 0=no symptoms, 4=inability to fall asleep at night due to symptoms) and afternoon (a 0-5 scale, with 0=no symptoms, 5=severe symptoms, unable to work or perform daily activities).
Incidence of Adverse events (AEs) | 32 weeks
  Incidence of AEs, including any abnormal physical examinations, abnormal vital signs, abnormal ECG, and abnormal lab testing.
Trough concentration at steady-state of CM310 | 32 weeks
  To evaluate the trough concentration at steady-state of CM310 for each dose group. Population pharmacokinetic analysis is performed using a nonlinear mixed-effects model.
Human thymus and activation-regulated chemokine (TARC) | 32 weeks
  Change from baseline in TARC at each evaluation time point for each dose group.
Fractional exhaled nitric oxide (FeNO). | 32 weeks
  Change from baseline in FeNO at each evaluation time point for each dose group.
Total IgE (immunoglobulin E) | 32 weeks
  Change from baseline in total IgE at each evaluation time point for each dose group.
Anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs). | 32 weeks
  Incidence of anti-drug antibodies (ADAs) and neutralizing antibodies (Nabs) (if applicable).

CONTACTS AND LOCATIONS:
Locations (1):
- China-Japan Friendship Hospital, Beijing, China